CLINICAL TRIAL: NCT00918411
Title: Post-marketing Clinical Study of Ramosetron Hydrochloride (Irribow Tablets) - A Preliminary Study to Evaluate the Co-primary Endpoint in Patients (Male) With Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: A Preliminary Study to Explore Clinical Endpoints in Patients (Male) With Diarrhea-predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 060-CL-500
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: diarrhea; IBS; Colonic diseases; YM060
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Colonic Diseases | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramosetron group (Experimental): oral
  Interventions: Drug: Ramosetron
- Placebo group (Placebo Comparator): oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramosetron — oral
  Other Names: Irribow; YM060
  Arms: Ramosetron group
Drug: Placebo — oral
  Arms: Placebo group

SUMMARY:
The purpose of this study is to explore and examine endpoints that allow evaluation of the "clinically significant improvements, focusing on the patient's chief complaint and the severity of major IBS symptoms" by this drug in patients with diarrhea-predominant irritable bowel syndrome (IBS).

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the Rome III Diagnostic Criteria
* Loose (mushy) or watery stools within the last 3 months

Exclusion Criteria:

* Patients having hyperthyroidism or hypothyroidism

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
IBS severity index (Japanese version) | 12 weeks

SECONDARY OUTCOMES:
Patient reported global assessment of relief of IBS symptoms | 12 weeks
Patient reported assessment of relief of abdominal discomfort and/or pain | 12 weeks
Patient reported assessment of improvement of abdominal bowel habits | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu

REFERENCES:
- [Derived] Ida M, Nishida A, Akiho H, Nakashima Y, Matsueda K, Fukudo S. Randomized, placebo-controlled, phase IV pilot study of ramosetron to evaluate the co-primary end points in male patients with irritable bowel syndrome with diarrhea. Biopsychosoc Med. 2017 Mar 16;11:8. doi: 10.1186/s13030-017-0093-9. eCollection 2017. PMID 28331539
- [Derived] Ida M, Nishida A, Akiho H, Nakashima Y, Matsueda K, Fukudo S. Evaluation of the irritable bowel syndrome severity index in Japanese male patients with irritable bowel syndrome with diarrhea. Biopsychosoc Med. 2017 Mar 11;11:7. doi: 10.1186/s13030-017-0092-x. eCollection 2017. PMID 28293280
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=060-CL-500